CLINICAL TRIAL: NCT00853255
Title: Phase 1 Inpatient Study of the Safety and Immunogenicity of One Dose of Live Influenza A Vaccine H7N3 (6-2) AA ca Recombinant (A/Chicken/British Columbia/CN-6/2004 x A/Ann Arbor/6/60 ca), a Live Attenuated Virus Vaccine Candidate for Prevention of Avian Influenza H7N3 Infection in the Event of a Pandemic
Brief Title: Group Study of the Safety of and Immune Response to a Single Dose of Bird Flu Vaccine (H7N3) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIR 260; CIR 260
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Influenza; Virus Diseases
Keywords: Bird Flu
MeSH Terms: conditions — Influenza, Human; Virus Diseases; Influenza in Birds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Participants will receive 0.5 mL of vaccine intranasally via an Accuspray device (0.25 mL in each nostril)
  Interventions: Biological: Live Influenza A Vaccine H7N3 (6-2) AA ca Recombinant (A/chicken/British Columbia/CN-6/2004 x A/Ann Arbor/6/60 ca)

INTERVENTIONS:
Biological: Live Influenza A Vaccine H7N3 (6-2) AA ca Recombinant (A/chicken/British Columbia/CN-6/2004 x A/Ann Arbor/6/60 ca) — Vaccine administered by nasal spray

SUMMARY:
Over the past decade, avian influenza (AI) has become a major health concern. The development of safe and effective vaccines against avian strains that infect people is important. The purpose of this study is to determine the safety of and immune response of an investigational AI vaccine in healthy adults against the H7N3 strain of avian influenza.

DETAILED DESCRIPTION:
The current pandemic risk associated with avian influenza H7N3 infection is significant, as an increasing number of humans are infected. H7 influenza transmission usually occurs in humans when they are exposed through direct contact to infected poultry or surfaces and objects contaminated by infected poultry feces. A pandemic occurs when a new influenza subtype emerges that infects humans, causes serious illness, and spreads easily between humans. The development of a safe and effective vaccine is necessary. The purpose of this study is to evaluate the safety and immunogenicity of a one-dose administration of the live, attenuated AI virus vaccine, H7N3 (6-2) AA ca Recombinant (A/chicken/British Columbia/CN-6/2004 x A/Ann Arbor/6/60 ca).

This study will last approximately 180 days. Participation in this study includes one 12-day hospital stay in an isolation unit at the University of Rochester Vaccine Evaluation Isolation Unit at St. Mary's Hospital in Rochester, NY. All participants will receive one dose of vaccine in nasal spray form at study entry. Participants will be admitted to the isolation unit 2 days prior to vaccination. A targeted physical exam, vital signs measurement, and nasal wash will occur daily following each vaccination until discharge. Participants will be discharged after two consecutive nasal washes on or after Day 7 are negative. Blood and urine collection will occur at selected timepoints throughout the study. Follow-up outpatient visits will occur approximately at Days 28, 56, and 180. A nasal wash and adverse events evaluation will occur at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Available for the duration of the trial
* For females, willing to use acceptable forms of contraception for the duration of the study. More information on this criterion can be found in the protocol.

Exclusion Criteria:

* Clinically significant neurologic, heart, lung, liver, rheumatologic, autoimmune, or kidney disease
* Behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may affect study participation
* Previously enrolled in an H7N3 influenza vaccine trial or in any study of an avian influenza vaccine
* Seropositive to the H7N3 influenza A virus (serum hemagglutination inhibition [HI] titer greater than 1:8)
* Illegal drug use or dependency determined by urine test
* Medical, work, or family problems as a result of alcohol or illicit drug use within 12 months prior to study entry
* History of severe allergic reaction
* Allergy to oseltamivir
* Asthma or reactive airways disease within 2 years prior to study entry
* History of Guillain-Barre syndrome
* HIV-infected
* Hepatitis C virus infected
* Positive for hepatitis B surface antigen (HBsAg)
* Known immunodeficiency syndrome
* Use of corticosteroids or immunosuppressive drugs within 30 days prior to vaccination. Participants who have used topical corticosteroids are not excluded.
* Receipt of live vaccines within 4 weeks prior to study vaccination
* Receipt of killed vaccines within 2 weeks prior to study vaccination
* Absence of spleen
* Receipt of blood products within 6 months prior to study vaccination
* Current smoker unwilling to stop smoking for the duration of the study
* Have traveled to the Southern Hemisphere within 14 days prior to study vaccination
* Have traveled on a cruise ship within 14 days prior to study vaccination
* Work in the poultry industry within 14 days prior to or after study vaccination
* Other investigational vaccine or drug within 30 days prior to study vaccination
* Allergy to eggs or egg products
* Other condition that, in the opinion of the investigator, may interfere with the study
* Pregnant or breastfeeding

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related reactogenicity events | During inpatient stage
Area under the curve of nasal viral shedding | Days 2 through 9
Development of serum antibody assessed by either HAI or MN assays | Throughout study

SECONDARY OUTCOMES:
Number of participants infected with the recombinant vaccine candidate | Throughout study
T-cell mediated and innate immune responses against recombinant vaccine candidate | Throughout study
Development of serum bank for testing effectiveness of vaccine against future viruses | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: John Treanor, MD, Principal Investigator — Infectious Diseases Division, University of Rochester Medical Center
Locations (1):
- University of Rochester Vaccine Evaluation Isolation Unit, St. Mary's Hospital, Rochester, New York, United States

REFERENCES:
- [Background] Alexander DJ. Avian influenza viruses and human health. Dev Biol (Basel). 2006;124:77-84. PMID 16447497
- [Background] Joseph T, McAuliffe J, Lu B, Jin H, Kemble G, Subbarao K. Evaluation of replication and pathogenicity of avian influenza a H7 subtype viruses in a mouse model. J Virol. 2007 Oct;81(19):10558-66. doi: 10.1128/JVI.00970-07. Epub 2007 Jul 18. PMID 17634234
- [Background] Joseph T, McAuliffe J, Lu B, Vogel L, Swayne D, Jin H, Kemble G, Subbarao K. A live attenuated cold-adapted influenza A H7N3 virus vaccine provides protection against homologous and heterologous H7 viruses in mice and ferrets. Virology. 2008 Aug 15;378(1):123-32. doi: 10.1016/j.virol.2008.05.021. Epub 2008 Jun 27. PMID 18585748
- [Background] Skowronski DM, Li Y, Tweed SA, Tam TW, Petric M, David ST, Marra F, Bastien N, Lee SW, Krajden M, Brunham RC. Protective measures and human antibody response during an avian influenza H7N3 outbreak in poultry in British Columbia, Canada. CMAJ. 2007 Jan 2;176(1):47-53. doi: 10.1503/cmaj.060204. PMID 17200390